CLINICAL TRIAL: NCT06427473
Title: Effectiveness of a Combined Diet and Mindfulness Program on Weight Loss in Breast Cancer Survivors: A Randomized Controlled Trial
Brief Title: Effectiveness of a Combined Diet and Mindfulness Program on Weight Loss in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, I-Ching Hou, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NYCU113018AE
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Weight Loss
Keywords: weight management; breast cancer survivors; mindfulness; Food Frequency Questionnaire
MeSH Terms: conditions — Breast Neoplasms; Weight Loss | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEM model (Experimental): subjects participate diet, exercise and mindfulness programs
  Interventions: Behavioral: Dietary program; Behavioral: Exercise program; Behavioral: Mindfulness program
- DE model (Active Comparator): subjects participate diet and exercise programs
  Interventions: Behavioral: Dietary program; Behavioral: Exercise program

INTERVENTIONS:
Behavioral: Dietary program — Participants will attend 8-week online dietary course. In addition to weekly classes, participants are required to photograph each meal.
Behavioral: Exercise program — Everyday walking steps more than 4000 steps. To accurately track participants' daily step counts, the research team provided quailfied pedometers.
Behavioral: Mindfulness program — Participants will attend 8-week online mindfulness course. In addition to weekly classes, participants practiced mindfulness individually for 5 minutes each day and maintained a mindfulness diary.
  Arms: DEM model

SUMMARY:
The study addresses the pressing issue of overweight and obesity among breast cancer patients, which exacerbates recurrence rates and mortality risks. Its primary objective is to assess the efficacy of two intervention models, the Diet, Exercise, and Mindfulness (DEM) model and the Diet and Exercise (DE) model, in facilitating weight loss, enhancing self-efficacy, mindfulness, and quality of life. The anticipated outcomes include long-term engagement in online self-learning, overcoming the limitations of ineffective self-management learning, and empowering healthcare professionals with scenario-based teaching materials. Through online platforms, patients can learn and review without constraints, ultimately achieving a holistic balance among physical, mental, and spiritual health.

DETAILED DESCRIPTION:
[Research Background] Breast cancer ranks first among cancers in women worldwide, with overweight and obesity being one of the high-risk factors for breast cancer. Moreover, overweight individuals within the breast cancer patient population also face higher recurrence rates and mortality risks. Assisting overweight or obese breast cancer women in weight loss to promote their well-being was the initial idea behind this study. The most common weight loss strategies include dietary management and regular exercise. In recent years, more studies have shown that effective weight loss also requires psychological interventions. Therefore, this study will combine dietary, exercise, and mindfulness-related interventions to assist breast cancer patients in more effective weight management.

[Research Objectives] To compare the effectiveness of two intervention measures, the Diet, Exercise, and Mindfulness (DEM) model and the Diet and Exercise (DE) model, on weight loss, self-efficacy, mindfulness tendency, and quality of life.

[Research Method] The study will involve a quantitative study, which plans to carry out a randomized controlled trial (RCT). This trial will compare the effects of two intervention measures, the DEM model and the DE model, on weight loss, self-efficacy, mindfulness tendency, and quality of life.

[Expected Results] Through the intervention provided by this study, patients can engage in long-term online self-learning and supplementary learning after returning home, reducing the limitations of ineffective self-management learning caused by negative emotions, treatment side effects, and sequelae in the early stages of cancer. Healthcare professionals can also use scenario-based teaching materials produced by this study to guide breast cancer survivors with ineffective weight self-management skills in practicing the necessary skills. Additionally, through online learning, patients can learn and review without pressure, saving time on transportation, easing carbon foot print and relearning effective weight management skills; even if they have faced major life threats in the past, they can turn adversity into blessings, achieving a balance among physical, mental, and spiritual health.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III breast cancer and completed treatment
* Body mass index (BMI) is greater than or equal to 24 kg/m2
* possess a smartphone

Exclusion Criteria:

* Pregnant or planning to become pregnant within six months
* Those who are unable to walk

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Physiological indicator I | baseline, 8 weeks, 24 weeks, 48 weeks
  BMI in kg/m2 (weight in kilograms divided by height in meters squared)
Physiological indicator II | baseline, 8 weeks, 24 weeks, 48 weeks
  Waist circumference in centimeter
Physiological indicator III | baseline, 8 weeks, 24 weeks, 48 weeks
  Body fat in percentage
Physiological indicator IV | baseline, 8 weeks, 24 weeks, 48 weeks
  Muscle mass in kilograms
Food Intake Frequency | baseline, 8 weeks, 24 weeks, 48 weeks
  Food Frequency Questionnaire
Mindful Awareness Attention | baseline, 8 weeks, 24 weeks, 48 weeks
  The minimum value is 1 and maximum value is 6, and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Weight Efficacy Lifestyle Questionnaire | baseline, 8 weeks, 24 weeks, 48 weeks
  The minimum value is 0 and maximum value is 10, and higher scores mean a better outcome.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | baseline, 8 weeks, 24 weeks, 48 weeks
  1. Item 1 to 28 the minimum value is 1 and maximum value is 4, and lower scores mean a better outcome.
  2. Item 29 to 30 the minimum value is 1 and maximum value is 7, and higher scores mean a better outcome.
Breast Cancer-Specific Quality of Life Questionnaire | baseline, 8 weeks, 24 weeks, 48 weeks
  The minimum value is 1 and maximum value is 4, and lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No